CLINICAL TRIAL: NCT05121194
Title: Adaptation and Evaluation of Virtual Group-Based Cognitive Behavior Therapy Classes for Mental Wellness in Public Safety Personnel
Brief Title: Evaluation of Virtual CBTm for Public Safety Personnel
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Shay-Lee Bolton, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H2021:196; PJI-175442 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2021-09-15; First posted 2021-11-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Cognitive Behaviour Therapy
Keywords: Mental Health; Telemedicine; Public Safety Personnel; Resiliency; Cognitive Behaviour Therapy; Evaluation; Intervention; Prevention
MeSH Terms: conditions — Psychological Well-Being | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ZOOM Video Conference Participants (Active Comparator): Participants will be offered the opportunity to join one of two weekly meeting times. Participants will be sent a link to join a Zoom videoconference session at the outset of each week, allowing them to log in at their chosen timeslot. These meeting times will be arranged based on discussions with the PAC around optimal timeslots for their shift workers. Sessions will be 90 minutes in length and will be facilitated by a minimum of 2 trained clinician facilitators and 1 research assistant. The session will include a PowerPoint presentation of the CBTm material in a lecture format. Participants will be invited and encouraged to discuss, comment and ask questions of the facilitators about the material throughout the presentation. Homework will be assigned each session relating to the material that was covered. Participants will have 1 week to work through and practice the skills learned, and this homework will be discussed at the next session.
  Interventions: Behavioral: Cognitive Behaviour Therapy
- WEB Online CBTm Course Participants (Active Comparator): Participants will receive access to the online self-guided CBTm course. The material is identical to the material taught in the facilitator-led group. Participants will receive access to the Class 1 upon joining the study at which point they can move through the material. The material is presented in a slide show format with pre-recorded audio to accompany each slide, in accordance with the material covered for in person classes. Material may be completed in a single sitting or they can choose to pause and return to it at a later time. Homework will be assigned as in Arm 1, through online forms at the end of each class. If a participant has questions, they can use a 'contact us' button, allowing questions to be sent to our research team. One week after completion of Class 1, participants will receive access to Class 2. The one-week timeframe prior to accessing the next class is used to mirror the timeline in the facilitator-led groups (Arm 1)
  Interventions: Behavioral: Cognitive Behaviour Therapy
- WAIT participants (No Intervention): (WAIT) participants will be assigned to a waitlist control. These individuals will not receive any type of active intervention but will continue to receive mental health questionnaires to complete in line with the ZOOM and WEB participants at weekly intervals. These individuals will be offered a choice of videoconference CBTm or online CBTm at completion of their waitlist period (6 months).

INTERVENTIONS:
Behavioral: Cognitive Behaviour Therapy — Group-based cognitive behaviour therapy (CBT) is an evidence-based treatment that allows service providers to interact with high volumes of individuals who need mental health support. CBT is the most well-researched and well-recognized of all psychotherapies, and is often considered the gold-standard in psychotherapy treatment. While CBT has shown efficacy in the treatment of a range of mental and substance use disorders, it has also been shown to be useful in building resiliency, being used as a tool to better cope during stressful life situations even among individuals who do not have an existing mental illness. Furthermore, research suggests that gains achieved in mental health during CBT are maintained long after treatment completion.
  Arms: WEB Online CBTm Course Participants; ZOOM Video Conference Participants

SUMMARY:
The principal aim of this study is to evaluate whether virtual CBTm is effective in improving mental wellness among public safety personnel (PSP). The investigators have adapted the CBTm classes to two virtual formats: 1) a facilitator-led set of virtual CBTm classes, and 2) an online self-guided version of the program.

Primary Objective: Can virtual CBTm increase resiliency among PSP?

Secondary Objectives:

i. Does virtual CBTm improve clinical symptoms of mental and substance use disorders (e.g., depression, anxiety, PTSD, alcohol abuse) among PSP? ii. Does virtual CBTm improve self-perceived health-related quality of life among PSP? iii. Does virtual CBTm reduce burnout among PSP?

Evaluation of all primary and secondary objectives will focus on clinically significant improvement in scores on well-validated measures. Steps to evaluate these objectives will include: 1) Recruit a cohort of PSP; 2) Assess baseline levels of resiliency, mental health symptoms, substance use, level of burnout, and current health-related quality of life; 3) Randomize individuals to one of two intervention arms or a waitlist control group; 4) Deliver CBTm in 2 different virtual formats; 5) Evaluate whether scores over time are significantly improved among individuals in each of the virtual CBTm groups compared with the waitlist control group. Comparisons of similarities and differences between the two intervention arms will also be conducted, particularly in terms of feasibility, acceptability, and facilitators/barriers of the virtual format for participants. The investigators will identify the demographic/symptom profiles of those who benefit most from each virtual-based CBTm.

DETAILED DESCRIPTION:
The study will be a nonblinded three-arm randomized controlled trial evaluating the effectiveness of a 5-session CBTm program. Arm 1 will be a videoconference-based, facilitator-led, group CBTm course (ZOOM); Arm 2 will be a self-guided online web-based CBTm course (WEB); and Arm 3 will be a waitlist control group (WAIT).

The investigators initially developed a 4-session (90 min each) facilitator-led CBTm program. As part of their initial pilot work with this population, they created a Project Advisory Committee (PAC), formed of researchers and PSP stakeholders and leaders. Based on their discussions with the PAC, it was recommended that a fifth class be added that focused on responding to traumatic events and stress using a CBT approach along with safety planning for managing crisis situations. As such, the program was adapted to a 5-session model for use in PSP. Session topics are as follows:

Session 1. Mindfulness, Basics of Cognitive Therapy, Thought Records Session 2. Mindfulness, Basics of Behaviour Therapy, Exposure Therapy Session 3. Mindfulness, Healthy Activity, Sleep Hygiene Session 4. Mindfulness, Goal Setting, Assertiveness Session 5. Mindfulness, Dealing with Stress and Stressful Experiences, Wellness Planning

For the proposed study, Arm 1 (ZOOM) participants will be offered the opportunity to join one of 2-3 weekly meeting times. Participants will be sent a link to join a Zoom videoconference session at the outset of each week, allowing them to log in at their chosen time slot. These meeting times will be arranged based on discussions with the PAC around optimal time slots for their shift workers. Sessions will be 90 minutes in length and will be facilitated by a minimum of 2 trained clinician facilitators and 1 research assistant. The session will include a PowerPoint presentation of the CBTm material in a lecture format. Participants will be invited and encouraged to discuss, comment and ask questions of the facilitators about the material throughout the presentation. Homework will be assigned each session relating to the material that was covered. Participants will have 1 week to work through and practice the skills learned, and this homework will be discussed at the next session. Arm 2 (WEB) participants will receive access to the online self-guided CBTm course. The material within that program is identical to the material taught within the facilitator-led groups. Participants will receive access to the Session 1 material upon joining the study at which point they will be able to move through the material at their own pace. The material is presented in a slide show format with pre-recorded audio to accompany each slide, in accordance with the material that they would cover if the class was held in-person. Material may be completed in a single sitting or the participant can choose to pause the session and return to it at a later time. Homework will be assigned as in the ZOOM arm through online forms that appear at the end of each session. These forms will be able to be completed online at any point during or after the session. Handouts will be able to be printed if the participant would like to complete the homework on paper. If the participant has any questions, they will have access to a 'contact us' button which will allow questions to be sent to the research team. These emails will be accessed daily by the research team. Some questions may need to be forwarded on to facilitators or clinicians depending on the content. One week after completion of Session 1, participants will receive access to Session 2. This one-week timeframe prior to accessing the next session is used to mirror most closely the time in which participants in the facilitator-led groups will have to practice the skills learned each week before another class is held. The online CBTm course has been in development through Safeandcertified.com, a company with substantial experience in developing and delivering courses for workplace safety and the SafeWork initiative in Manitoba. Arm 3 (WAIT) participants will be assigned to a waitlist control. These individuals will not receive any type of active intervention but will continue to receive mental health questionnaires to complete in line with the ZOOM and WEB participants at weekly intervals. These individuals will be offered a choice of videoconference CBTm or online CBTm at completion of their waitlist period (6 months).

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be of legal adult status (age 18 or older)
* currently employed as a public safety worker (e.g., police officer, law enforcement, fire fighter, paramedic, dispatcher, correctional worker),
* and located within Manitoba

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in 10-item Connor-Davidson Resilience Scale | 5 weeks (change from baseline to end of treatment)
  changes in scores
  This 10-item version of the original 25-item scale was developed to measure resiliency.
  Scale Range: 0-40 (total score) Lower scores indicate less resiliency (i.e., worse outcome) Higher scores indicate more resiliency (i.e., better outcome)

SECONDARY OUTCOMES:
Change in 10-item Connor-Davidson Resilience Scale | 6 months (change from end of treatment to 6-month follow-up)
  changes in scores
  This 10-item version of the original 25-item scale was developed to measure resiliency.
  Scale Range: 0-40 (total score) Lower scores indicate less resiliency (i.e., worse outcome) Higher scores indicate more resiliency (i.e., better outcome)
Change in Short Form 12 (SF-12) | 5 weeks (change from baseline to end of treatment)
  change in scores
  This 12-item version of the original 36-item scale is a self-report of health-related quality of life. The scale includes 2 subscales, the physical component score (PCS-12) and mental component score (MCS-12) Scale Range: 0-100 (standard score for total and each subscale) Lower scores indicate worse physical and mental health functioning (i.e., worse outcome) Higher scores indicate better physical and mental health functioning (i.e., better outcome)
Change in Short Form 12 (SF-12) | 6 months (change from end of treatment to 6-month follow-up)
  change in scores
  This 12-item version of the original 36-item scale is a self-report of health-related quality of life. The scale includes 2 subscales, the physical component score (PCS-12) and mental component score (MCS-12) Scale Range: 0-100 (standard score for total and each subscale) Lower scores indicate worse physical and mental health functioning (i.e., worse outcome) Higher scores indicate better physical and mental health functioning (i.e., better outcome)
Change in Maslach Burnout Inventory-Human Services Survey (MBI-HSS) | 5 weeks (change from baseline to end of treatment)
  change in scores
  Designed specifically for assessing burnout among those working in the human services. The MBI-HSS comprises 22 questions across 3 subscales; Emotional Exhaustion (EE)-9 questions, Depersonalization (DP)-5 questions, and self-perceived lack of Personal Accomplishment (PA)-8 questions.
  Scale Range: EE (0-54), DP (0-30), PA (0-48) Lower scores indicate less EE, DP, and PA (i.e., better outcome) Higher scores indicate more EE, DP, and PA (i.e., worse outcome)
Change in Maslach Burnout Inventory-Human Services Survey (MBI-HSS) | 6 months (change from end of treatment to 6-month follow-up)
  change in scores
  Designed specifically for assessing burnout among those working in the human services. The MBI-HSS comprises 22 questions across 3 subscales; Emotional Exhaustion (EE)-9 questions, Depersonalization (DP)-5 questions, and self-perceived lack of Personal Accomplishment (PA)-8 questions.
  Scale Range: EE (0-54), DP (0-30), PA (0-48) Lower scores indicate less EE, DP, and PA (i.e., better outcome) Higher scores indicate more EE, DP, and PA (i.e., worse outcome)
Change in Patient Health Questionnaire 9-Item (PHQ-9) | 5 weeks (change from baseline to end of treatment)
  change in scores
  Validated and reliable 9-item measure for assessing the severity of depression in the general population Scale range: 0-27 (total score_ Lower scores indicate lower severity of depressive symptoms (i.e., better outcome) Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)
Change in Patient Health Questionnaire 9-Item (PHQ-9) | 6 months (change from end of treatment to 6-month follow-up)
  change in scores
  Validated and reliable 9-item measure for assessing the severity of depression in the general population Scale range: 0-27 (total score_ Lower scores indicate lower severity of depressive symptoms (i.e., better outcome) Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)
Change in Generalized Anxiety Disorder 7-Item (GAD-7) | 5 weeks (change from baseline to end of treatment)
  change in scores
  This 7-item measure assesses anxiety in the general population Scale range: 0-21 (total score) Lower scores indicate lower severity of anxiety symptoms (i.e., better outcome) Higher scores indicate higher severity of anxiety symptoms (i.e., worse outcome)
Change in Generalized Anxiety Disorder 7-Item (GAD-7) | 6 months (change from end of treatment to 6-month follow-up)
  change in scores
  This 7-item measure assesses anxiety in the general population Scale range: 0-21 (total score) Lower scores indicate lower severity of anxiety symptoms (i.e., better outcome) Higher scores indicate higher severity of anxiety symptoms (i.e., worse outcome)
Change in Alcohol Use Disorders Identification Test (AUDIT) | 5 weeks (change from baseline to end of treatment)
  change in scores
  This 10-item screening tool is used to assess alcohol consumption, drinking behaviors, and alcohol-related problems Scale range: (0-40) A score of 8 or more is associated with harmful or hazardous drinking, a score of 13 or more in women, and 15 or more in men, is likely to indicate alcohol dependence.
Change in Alcohol Use Disorders Identification Test (AUDIT) | 6 months (change from end of treatment to 6-month follow-up)
  change in scores
  This 10-item screening tool is used to assess alcohol consumption, drinking behaviors, and alcohol-related problems Scale range: (0-40) A score of 8 or more is associated with harmful or hazardous drinking, a score of 13 or more in women, and 15 or more in men, is likely to indicate alcohol dependence.
Change in Cannabis Use Disorders Identification Test (CUDIT-R) | 5 weeks (change from baseline to end of treatment)
  change in scores
  This 8-item screening tool was developed to assess possible cannabis use issues.
  Scale range: (0-32) Scores of 8 or more indicate hazardous cannabis use, while scores of 12 or more indicate a possible cannabis use disorder for which further intervention may be required.
Change in Cannabis Use Disorders Identification Test (CUDIT-R) | 6 months (change from end of treatment to 6-month follow-up)
  change in scores
  This 8-item screening tool was developed to assess possible cannabis use issues.
  Scale range: (0-32) Scores of 8 or more indicate hazardous cannabis use, while scores of 12 or more indicate a possible cannabis use disorder for which further intervention may be required.
Change in Five-Facet Mindfulness Questionnaire (FFMQ-15) | 5 weeks (change from baseline to end of treatment)
  change in scores
  This 15-item scale is used to assess level of mindfulness (observing, describing, etc).
  Scale range: (0-75) Lower scores indicate lower level of mindfulness (i.e., worse outcome) Higher scores indicate higher level of mindfulness (i.e., better outcome)
Change in Five-Facet Mindfulness Questionnaire (FFMQ-15) | 6 months (change from end of treatment to 6-month follow-up)
  change in scores
  This 15-item scale is used to assess level of mindfulness (observing, describing, etc).
  Scale range: (0-75) Lower scores indicate lower level of mindfulness (i.e., worse outcome) Higher scores indicate higher level of mindfulness (i.e., better outcome)
Change in The Posttraumatic Stress Disorder Checklist DSM-5 (PCL-5) | 5 weeks (change from baseline to end of treatment)
  change in scores
  This questionnaire is a 20-item self-report measure of posttraumatic stress disorder Scale range: 0-80 (total score) Lower scores indicate lower severity of PTSD symptoms (i.e., better outcome) Higher scores indicate higher severity of PTSD symptoms (i.e., worse outcome)
Change in The Posttraumatic Stress Disorder Checklist DSM-5 (PCL-5) | 6 months (change from end of treatment to 6-month follow-up)
  change in scores
  This questionnaire is a 20-item self-report measure of posttraumatic stress disorder Scale range: 0-80 (total score) Lower scores indicate lower severity of PTSD symptoms (i.e., better outcome) Higher scores indicate higher severity of PTSD symptoms (i.e., worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Shay-Lee Bolton, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No